CLINICAL TRIAL: NCT01771926
Title: Lifestyle Modification and Potato Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFHNRC024
Record Dates: First submitted 2012-03-29; First posted 2013-01-18 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: resistant starch; lifestyle intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Resistant Starch Potatoes (Experimental): Subjects will receive 1 serving daily for 8 weeks during the weight loss group sessions.
  Interventions: Other: potatoes
- Low Resistant Starch Potatoes (Experimental): Subjects will receive 1 serving daily for 8 weeks during the weight loss group sessions.
  Interventions: Other: potatoes
- Other Carbohydrate Source (Placebo Comparator): Subjects will receive 1 serving daily for 8 weeks during the weight loss group sessions.
  Interventions: Other: other carbohydrate

INTERVENTIONS:
Other: potatoes — Daily intake of assigned treatment for 8 weeks
  Arms: High Resistant Starch Potatoes; Low Resistant Starch Potatoes
Other: other carbohydrate — Daily intake of assigned treatment for 8 weeks
  Arms: Other Carbohydrate Source

SUMMARY:
The investigators hypothesize that consumption of potatoes is a healthy adjunct to lifestyle intervention in overweight and obese glucose intolerant adults. We will evaluate the effects of the consumption of potatoes (high or low resistant starch) vs. commonly consumed carbohydrate sources on glucose tolerance; and ( the extent to which potato consumption alters markers of lipid metabolism and inflammation in the context of a lifestyle intervention program.

DETAILED DESCRIPTION:
Our primary objective is to compare the effects of potato consumption to those of commonly consumed carbohydrate sources on glucose tolerance and other cardiometabolic risk factors in overweight and obese, glucose intolerant men and women participating in a lifestyle intervention program. We hypothesize that consumption of potatoes is a healthy adjunct to lifestyle intervention in overweight and obese glucose intolerant adults. Our specific aims include: (1) to evaluate of the effects of the consumption of potatoes (high or low resistant starch) vs. commonly consumed carbohydrate sources on glucose tolerance; and (2) to determine the extent to which potato consumption alters markers of lipid metabolism and inflammation in the context of a lifestyle intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20-65 years of age.
* Overweight or obese (BMI 25 - 39.9 Kg/m2)
* Impaired Glucose Tolerance: fasting glucose between 100-125 mg/dL
* Willingness to comply with the demands of the experimental protocol
* Sedentary lifestyle

Exclusion Criteria

* Major medical condition
* Smokers
* Unable to perform moderate exercise
* Use of medications that alter glucose or lipid metabolism
* Pregnant or lactating

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Glucose Tolerance | Days 0, 14, 28, 42, 56

SECONDARY OUTCOMES:
Weight Loss | Days 0, 14, 28, 42, 56
Functional Fitness | Days 0 and 57

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Raatz, PhD, MPH, RD, Principal Investigator — USDA GFHNRC
Locations (1):
- Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center — http://www.ars.usda.gov/main/site_main.htm?modecode=54-50-00-00